CLINICAL TRIAL: NCT00005367
Title: Epidemiology of Long QTand Asian Sudden Death in Sleep
Status: Completed | Type: Observational
Sponsor: Utah State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4254; R01HL049432 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Arrhythmia; Death, Sudden, Cardiac; Long QT Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To conduct a cross-sectional epidemiologic study of the determinants of prolonged heart rate corrected QT interval (QTc) among 300 men and 300 woman in the population with the highest known risk of SUDS: Southeast Asian refugees in Thailand. .

DETAILED DESCRIPTION:
BACKGROUND:

Sudden and unexplained death in sleep (SUDS) is a leading cause of death of young men in several Asian populations. The immediate cause is ventricular fibrillation in the absence of known disease. A strong environmental component may be inferred from the regional nature of SUDS in groups that are culturally and genetically distinct and the rapid decline in rates of SUDS after migration of Southeast (SE) Asian refugees to the United States. Risk of SUDS rises sharply to a peak among men aged 35 years of age, then declines with increasing age. In a pilot studies of SE Asian refugee men in Thailand with the highest known risk of SUDS, the investigators documented high-prevalences of prolonged heart rate corrected QT interval (QTc), thiamine deficiency, hypokalemia, and a positive association between poor thiamine status, measured by erythrocyte transketolase activity (ETK), and QTc. These limited studies were unable to precisely quantify the relationship between QTc and thiamine status, lacked sufficient power to examine the relationship between QTc and hypokalemia, did not include other electrolytes, and did not address the striking differences in risk of SUDS by sex and age.

DESIGN NARRATIVE:

The study was cross-sectional in design. During a 14-month period, informed consent was obtained from subjects selected in an age-stratified random sample of refugees scheduled for routine medical screening. Blood samples, 12-lead and 24-hour ECGs, and interview data were collected to test the following hypotheses: (1) mean QTc was greater in men than women, (2) mean QTc was greater in men aged 30-39 years than in men younger or older; no similar relationship was expected among women, (3) QTc was positively correlated with poor thiamine status, measured by erythrocyte transketolase activity, (4-6) QTc was negatively correlated with serum levels of potassium, magnesium, and total calcium, and (7) QTc was associated with abnormalities of autonomic control of the heart, as indicated by power spectral analysis of heart rate variability. Secondary aims included studying interactions of thiamine status and electrolytes in the prolongation of QTc, dynamic analysis of QT variation by heart rate level in 24-hr ECGs, and collection of blood specimens for later genetic studies

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-02; Study Completion 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Munger — Utah State University

REFERENCES:
- [Background] Munger RG, Booton EA. Bangungut in Manila: sudden and unexplained death in sleep of adult Filipinos. Int J Epidemiol. 1998 Aug;27(4):677-84. doi: 10.1093/ije/27.4.677. PMID 9758125